CLINICAL TRIAL: NCT06456034
Title: Testing a Perinatal Palliative Care Intervention Program Within Standard Perinatal Healthcare: Pilot Testing Protocol
Brief Title: Pilot-testing a Perinatal Palliative Care Intervention Program
Acronym: PPC-pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Laure Dombrecht, Postdoctoral researcher, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PPC-pilot
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Perinatal Palliative Care; Life-limiting Fetal Diagnosis; Life-limiting Neonatal Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline group (No Intervention): Receives care as usual after severe perinatal diagnosis
- Perinatal palliative care group (Experimental): Receives a new perinatal palliative care intervention after severe perinatal diagnosis
  Interventions: Behavioral: Perinatal palliative care

INTERVENTIONS:
Behavioral: Perinatal palliative care — Intervention group will receive specialized perinatal palliative care support from moment of severe perinatal diagnosis. This intervention is aimed at 5 major care components, namely 1. Support offered by a fixed perinatal palliative care team, 2. that team has received specialized perinatal palliative care training, 3. care is structured within a new perinatal palliative care approach or pathway, including fixed means of communication with team members, 4. psychological support is structurally being offered to parents and healthcare providers, and 5. debriefings after every perinatal death are being organized in the involved team.
  Arms: Perinatal palliative care group

SUMMARY:
The objective of this pilot trial is to implement a new perinatal palliative care intervention program tailored to the Flemish context, which aims to provide care to parents who receive a severe foetal/neonatal diagnosis for their (unborn) child and to their healthcare providers. Additionally, we aim to evaluate the feasibility and preliminary effectiveness by comparing measured variables to the baseline measurement done in the same hospital wards beforehand.

ELIGIBILITY:
Inclusion Criteria:

* Parents:

  * who receive a severe foetal diagnosis for their unborn child and decide to continue the pregnancy after 20 weeks of gestation , or
  * who receive a severe foetal diagnosis for their unborn child after 20 weeks gestation and decide to terminate the pregnancy (with or without feticide) resulting in the stillbirth of their child
* Parents who receive a severe neonatal diagnosis for their live-born infant in the first week after birth

Additional inclusion criteria for parents:

* Parents are either Dutch speaking, or are willing to participate with support from a (phone or real life) interpreter, in collaboration with the "Agentschap Integratie & Inburgering"
* Parents are older than 18
* Parents are not suffering from an officially diagnosed psychiatric disorder prior to receiving the severe diagnosis of their child
* Parents are deemed (emotionally) approachable for the current study by the treating physician

For each family included in the pilot study, the physicians and nurses/midwives who will be/are most closely involved in the care of the infant and the parents will also be asked to participate. If healthcare providers refuse to provide informed consent to participate in the study, their data will be deemed as missing for that case (parental outcomes are considered as the primary outcome measures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
NeoComfort scale | every four hours (six times per day) during care provision for neonates only
  The validated NeoComfort scale will be used to assess pain and discomfort. The COMFORTneo scale is composed of 7 behavioral dimensions: As respiratory response applies to ventilated neonates only, and crying to spontaneously breathing neonates only (including those requiring continuous positive airway pressure), the rater will actually rate 6 dimensions. Alertness, calmness/agitation, facial tension, muscle tone, body movement are rated for all neonates. As responses are on a 1 to 5 Likert scale, total scores range from 6 to 30-with higher scores indicating more pain.scores range from 6 to 30-with higher scores indicating more pain.
Administered medication and procedures | during care provision
  All medication administration and procedures followed are registered throughout the care trajectory. Duration or timing is impossible to predict.
Contact moments with healthcare providers | during care provision
  Contact moments between healthcare providers and parents are registered throughout the care trajectory. Duration or timing is impossible to predict.
Parental Perinatal Grief Scale | 2 weeks after final contact moment or 6 months post inclusion
  Scoring of the parental Perinatal Grief Scale. The short version of the Perinatal Grief Scale consists of 33 items that represents three subscales each consisting of 11 items: active grief (sadness, missing the baby, crying for the baby), difficulty coping (difficulty in dealing with normal activities with other people, withdrawal and depression), and despair (feelings of worthlessness and hopelessness). Each item is scored on a 5-point likert scale, resulting in a possible range of 33-165. Higher scores reflect more intense grief.
Parental Brief-COPE | 2 weeks after final contact moment or 6 months post inclusion
  Scoring of parental Brief-COPE (Coping Orientation to Problems Experienced Inventory) questionnaire. The Brief-COPE is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. "Coping" is defined broadly as an effort used to minimize distress associated with negative life experiences. The scale can determine someone's primary coping styles with scores on the following three subscale: Problem-Focused Coping; Emotion-Focused Coping; and Avoidant Coping. Scores are presented for the three overarching coping styles as average scores (sum of item scores divided by number of items), indicating the degree to which the respondent has been engaging in that coping style (higher scores = more engagement of that coping style).
Parental Satisfaction of Perinatal Palliative Care | 2 weeks after final contact moment or 6 months post inclusion
  Scoring of The Parental Satisfaction of Perinatal Palliative Care Instrument, which was developed to identify and measure parental satisfaction in perinatal palliative care for parents who opt to continue a pregnancy with a life-limiting fetal diagnosis. The instrument measures parent-reported care delivery addressing the pregnancy time continuum in three scales (Prenatal; Intrapartum; Postnatal). Items in the instrument are on a Likert scale from 1-7, with 1 indicating "strongly disagree," 4 indicating "does not apply/neutral," and 7 indicating "strongly agree." Higher scores reflect higher parental perception of quality care delivery. The Prenatal Scale includes 37 items (range from 37-259); the Intrapartum Scale includes 37 items (range from 37-259); and the Postnatal Scale includes 44 items (range from 44-308).
Healthcare provider Compassion Satisfaction and Fatigue questionnaire | 2 weeks after final contact moment or 6 months post inclusion
  Scoring of Healthcare provider Compassion Satisfaction and Fatigue questionnaire. ProQOL is a survey consisting of 30 items scaled on a five-point Likert scale, measuring three subscales consisting of 10 items each: Compassion Satisfaction, Burnout and Secondary Traumatic Stress. The Compassion satisfaction scale is about the pleasure derived from your work, with higher scores indicating that you derive a good deal of professional satisfaction from your position (range of 10-50). The burnout subscale is associated with feelings of hopelessness and difficulties in dealing with work or in doing your job effectively. Higher scores on this scale mean that you are at higher risk for burnout (range of 10-50). The secondary traumatic stress scale is about your work-related, secondary exposure to extremely or traumatically stressful events, with a higher score indicating a higher amount of experienced secondary traumatic stress (range of 10-50).
Healthcare provider Professional Satisfaction with Provided Care | 2 weeks after final contact moment or 6 months post inclusion
  Scoring of Healthcare provider Professional Satisfaction with Provided Care. This is a self-developed (not yet validated) questionnaire on Professional Satisfaction with Provided Care consisting of 48 items, based on the existing Parental Satisfaction of Perinatal Palliative Care Instrument used in the parental assessment, to assess whether healthcare providers are satisfied with the perinatal palliative care they and their team provided in a particular case, including satisfaction with communication among the team, and communication with parents. Psychometric properties of the scale need to be determined after the pilot test.
Healthcare provider experienced (psychological) support | 2 weeks after final contact moment or 6 months post inclusion
  Scoring of Healthcare provider experienced (psychological) support. This is a short, self-developed (not yet validated) questionnaire consisting of 6 items for physicians or 6 items for nurses, to assess the amound of (psychological) support that healthcare providers received during the care provision for this particular case. Psychometric properties of the scale need to be determined after the pilot test.

SECONDARY OUTCOMES:
Parental feasibility and acceptability of pilot | 2 weeks after final contact moment or 6 months post inclusion
  Parental feasibility and acceptability of pilot. As assessed by means of interviews.
Healthcare provider feasibility and acceptability of pilot | 2 weeks after final contact moment or 6 months post inclusion
  Healthcare provider feasibility and acceptability of pilot. As assessed by means of interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Cools, Principal Investigator — Brussels University Hospital; Kristien Roelens, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - UZ Brussels, Brussels
  - UZ Gent, Ghent

IPD SHARING:
Plan to Share IPD: No